CLINICAL TRIAL: NCT00509925
Title: A 32-week National, Single-centre, Open-labelled, Randomised, Crossover Trial Comparing Energy Expenditure With Insulin Detemir Versus NPH Insulin Using a Basal-Bolus Regimen With Insulin Aspart as Mealtime Insulin in Subjects With Type 1 Diabetes
Brief Title: Effect of Insulin Detemir on Use of Energy in Type 1 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1761; 2006-003060-59 (EudraCT Number)
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental): Insulin detemir for 16 weeks (treatment period 1) followed by insulin NPH treatment for 16 weeks (treatment period 2) in addition to meal-time insulin aspart
  Interventions: Drug: insulin detemir; Drug: insulin NPH; Drug: insulin aspart
- Treatment period 2 (Experimental): Insulin NPH for 16 weeks (treatment period 1) followed by insulin detemir treatment for 16 weeks (treatment period 2) in addition to meal-time insulin aspart
  Interventions: Drug: insulin detemir; Drug: insulin NPH; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target dose tritation (dose adjusted individually), s.c. (under the skin) injection
Drug: insulin NPH — Treat-to-target dose tritation (dose adjusted individually), s.c. (under the skin) injection
Drug: insulin aspart — Treat-to-target dose tritation (dose adjusted individually), s.c. (under the skin) injection

SUMMARY:
This trial is conducted in Europe. The purpose of this trial is to investigate if there is any change in the mechanism of energy expenditure (i.e. the way in which energy is used) in patients with type 1 diabetes, whilst taking two different, commercially available insulins for the treatment of their diabetes.

DETAILED DESCRIPTION:
The study had been temporarily halted due to an unplanned interim analysis. The Sponsor is now aware that a further interim analysis has been performed by the site and therefore a decision has been made not to recommence the study

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than 12 months
* Current treatment: Basal-bolus insulin regimen for more than three months (i.e. at least one daily injection of long-acting insulin (including insulin glargine) and fast-acting insulin with each main meal)
* HbA1c (glycosylated haemoglobin A1c) between 7.0 and 11.0%
* Able and willing to maintain consistent physical activity level throughout the entire study period
* Able and willing to maintain consistent eating habits throughout the entire study period

Exclusion Criteria:

* Proliferative retinopathy that has required acute treatment within the last six months
* Recurrent major hypoglycaemia or hypoglycaemic unawareness as judged by the Investigator
* Liver, kidney or heart problems as judged by the Investigator
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures
* Known or suspected allergy to trial products or related products
* Receipt of any investigational drug within one month prior to this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Guildford, United Kingdom

REFERENCES:
- [Result] Zachariah S, Sheldon B, Shojaee-Moradie F, Jackson NC, Backhouse K, Johnsen S, Jones RH, Umpleby AM, Russell-Jones DL. Insulin detemir reduces weight gain as a result of reduced food intake in patients with type 1 diabetes. Diabetes Care. 2011 Jul;34(7):1487-91. doi: 10.2337/dc11-0098. Epub 2011 May 18. PMID 21593292
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One single site in United Kingdom.
Pre-assignment Details: Eligible subjects were those with type 1 diabetes treated with insulin for at least 3 months having a body mass index (BMI) of 40.0 kg/m2 at most and a glycosylated haemoglobin A1c (HbA1c) between 7-11% qualifying for an intensified insulin treatment based on the treat-to-target concept. The randomisation target for this study was 30 subjects.
Groups:
- Insulin Detemir First, Then Insulin NPH: Insulin detemir + insulin aspart once or twice daily for 16 weeks (treatment period 1) followed by switch to insulin NPH + insulin aspart (dose adjusted individually) once or twice daily for 16 weeks (treatment period 2)
- Insulin NPH First, Then Insulin Detemir: Insulin NPH + insulin aspart (dose adjusted individually) once or twice daily for 16 weeks (treatment period 1) followed by switch to insulin detemir + insulin aspart (dose adjusted individually) once or twice daily for 16 weeks (treatment period 2)
Period: Overall Study
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Personal reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Trial Population: The entire trial population includes groups randomised to receive either insulin detemir or insulin NPH as their first treatment.
Arm/Group | Entire Trial Population
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 28.0 (3.6)
Body composition: Fat Mass [Mean (Standard Deviation); unit: kg] | 21.3 (9.3)
Body composition: Lean Body Mass [Mean (Standard Deviation); unit: kg] | 60.6 (10.8)
FPG [Mean (Standard Deviation); unit: mmol/L] — Fasting plasma glucose
  mmol/L | 10.4 (3.6)
HbA1c [Mean (Standard Deviation); unit: percentage of total haemoglobin] — Glycosylated haemoglobin A1c (HbA1c)
  percentage of total haemoglobin | 8.2 (1.0)
Height [Mean (Standard Deviation); unit: meters] | 1.7 (0.1)
Waist:hip ratio [Mean (Standard Deviation); unit: percentage of hip circumference] — Waist:hip ratio was calculated as waist average in cm divided by hip average in cm, and multiplied by 100.
  percentage of hip circumference | 93.5 (7.5)
Weight [Mean (Standard Deviation); unit: kg] | 81.9 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Total Energy Expenditure, Double-labelled Water Method
Description: Total energy expenditure (TEE) measured after each treatment period by the double-labelled water (DLW) method. This technique required subjects to label their body water using oral administration of water labelled with 2 stable isotopes (2H218O). The clearance of 2H and 18O was measured over a two week period with daily collections of urine. The difference between the clearance of 2H and 18O is a measure of CO2 production rate. This can be converted to provide a measure of energy expenditure.
Time Frame: Weeks 14-16, weeks 30-32
Population: The analysis was performed on an ITT (Intent-to-Treat) analysis set. The ITT analysis set consisted of all subjects who received at least one post-treatment value of the primary endpoint.
Measure: Mean (Standard Deviation); unit: kcal/day
Groups:
- Insulin Detemir: Insulin detemir + insulin aspart (dose adjusted individually) once or twice daily in either the 1st or 2nd intervention period
- Insulin NPH: Insulin NPH + insulin aspart (dose adjusted individually) once or twice daily in either the 1st or 2nd intervention period
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 13 | 13
kcal/day | 2942.2 (683.9) | 3007.2 (649.9)

2. Secondary Outcome: Component of Total Energy Expenditure: Resting Energy Expenditure (REE)
Description: Resting energy expenditure (REE) is a component of TEE (total energy expenditure). It was measured at 2 different timepoints during the trial using indirect calorimetry (measurement of O2 consumption/CO2 production) after an overnight fast when subjects would be metabolising a mixture of carbohydrate and free fatty acid. This technique allowed the calculation of the rate of carbohydrate and lipid oxidation.
Time Frame: Week 14, week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 22
kcal/day | 1932.5 (443.5) | 2034.5 (368.7)

3. Secondary Outcome: Component of Total Energy Expenditure: Diet Induced Thermogenesis (DIT)
Description: Diet induced thermogenesis (DIT) is a component of TEE (total energy expenditure) and is the energy expenditure following feeding for anabolic processes. Subjects fasted overnight and rested for 1 hour. Multiple measurements of REE (resting energy expenditure) were taken. A fixed 600 kcal liquid meal was given and REE was measured over the next 3 hours. DIT was calculated as area under the curve of total REE-resting REE for the 3-hour period and was then converted to a per day measurement by taking into account each individual's average daily food intake.
Time Frame: Week 14, week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 21
kcal/day | 73.0 (33.9) | 74.3 (33.2)

4. Primary Outcome: Total Energy Expenditure, Dietary Record Method
Description: The total energy expenditure (TEE) measured after each treatment period by the dietary record method. The calculation of energy balance is accomplished by compiling an accurate record of food intake over a period of time and measuring any changes in body weight that occur during that time. Data from the 7-day food diary was used to calculate TEE.
Time Frame: Weeks 14-16, weeks 30-32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 21 | 21
kcal/day | 2017.9 (501.4) | 2181.0 (559.8)

5. Secondary Outcome: Component of Total Energy Expenditure: Physical Activity Thermogenesis
Description: Physical activity thermogenesis is a component of TEE (total energy expenditure). Subjects were asked not to change their physical activity levels. Physical activity thermogenesis can be calculated as the difference between TEE minus (REE + DIT), as long as volitional exercise is unchanged. Volitional exercise was assessed using Actiheart 3-D monitor readings. Subjects were asked to measure their normal activity for between 1 and 5 days prior to their visits at week 16 and week 32).
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 22 | 21
kcal/day | 588.5 (358.4) | 542.7 (281.6)

6. Secondary Outcome: Component of Total Energy Expenditure: Non-exercise Activity Thermogenesis (NEAT)
Description: Non-exercise activity thermogenesis is a component of TEE (total energy expenditure). Thermic efficiency was assessed by measuring O2 consumption/CO2 production while the subject exercised on a bike for 20 minutes while hooked up to a device that recorded their respiration (visit in week 14 and week 30). If thermic efficiency was unchanged and volitional exercise was unchanged, then any change in physical activity thermogenesis was due to changes in NEAT.
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 17 | 17
kcal/day | 1163.7 (1138.7) | 1170.0 (1084.6)

7. Secondary Outcome: Body Weight
Description: Body weight after each treatment period.
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Insulin Detemir First, Then Insulin NPH: Insulin detemir + insulin aspart (dose adjusted individually) once or twice daily for 16 weeks (treatment period 1) followed by switch to insulin NPH + insulin aspart (dose adjusted individually) once or twice daily for 16 weeks (treatment period 2)
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 22 | 22
kg
  Treatment period 1, N= 12, 10 | 80.6 (9.8) | 86.0 (11.7)
  Treatment period 2, N= 10, 12 | 82.9 (10.7) | 84.8 (11.6)

8. Secondary Outcome: Lean Body Mass
Description: Lean body mass was measured using Bioelectrical Impedance Analysis (BIA), a method used for estimating body composition.
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 21 | 22
kg
  Treatment period 1, N=12, 10 | 58.9 (9.9) | 63.7 (12.3)
  Treatment period 2, N=9, 12 | 59.9 (11.2) | 64.3 (12.0)

9. Secondary Outcome: Fat Mass
Description: Fat mass was measured using Bioelectrical Impedance Analysis (BIA), a method used for estimating body composition.
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 21 | 22
kg
  Treatment period 1, N=12, 10 | 21.7 (9.2) | 22.3 (10.8)
  Treatment period 2, N=9, 12 | 23.0 (8.5) | 19.2 (8.5)

10. Secondary Outcome: Waist:Hip Ratio
Description: At each time-point, 3 measurements each of waist and hip circumference were taken, then an average across the three measurements was calculated for both and the ratio was calculated as the waist average in cm divided by hip average in cm, and multiplied by 100.
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of hip circumference
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 22 | 22
percentage of hip circumference
  Treatment period 1, N= 12, 10 | 92.4 (9.3) | 94.4 (5.9)
  Treatment period 2, N= 10, 12 | 92.4 (9.4) | 94.8 (5.6)

11. Secondary Outcome: Hormonal Assessment: Adiponectin
Description: Adiponectin levels after each treatment period.
Time Frame: Week 14, week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 21 | 21
ng/ml
  Treatment period 1, N=12, 10 | 15978.3 (9108.9) | 11361.0 (3540.7)
  Treatment period 2, N=9, 11 | 15189.5 (10470.8) | 11053.3 (2956.1)

12. Secondary Outcome: Hormonal Assessment: Insulin-like Growth Factor-1
Description: Insulin-like growth factor-1 (IGF-1) levels after each treatment period.
Time Frame: Week 14, week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 21 | 19
ng/ml
  Treatment period 1, N=12, 9 | 212.3 (114.5) | 206.8 (112.2)
  Treatment period 2, N=9, 10 | 179.8 (76.4) | 168.4 (60.2)

13. Secondary Outcome: Hormonal Assessment: Resistin
Description: Resistin levels after each treatment period.
Time Frame: Week 14, week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 21 | 21
ng/ml
  Treatment period 1, N=12, 10 | 8.2 (2.4) | 10.2 (5.4)
  Treatment period 2, N=9, 11 | 8.4 (2.5) | 16.2 (13.2)

14. Secondary Outcome: Hormonal Assessment: Leptin
Description: Leptin levels after each treatment period.
Time Frame: Week 14, week 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 21 | 21
ng/ml
  Treatment period 1, N=12, 10 | 9.4 (7.0) | 10.5 (12.1)
  Treatment period 2, N=9, 11 | 9.9 (5.9) | 6.6 (7.7)

15. Secondary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Glycosylated haemoglobin A1c (HbA1c) after each treatment period.
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total haemoglobin
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 21 | 22
percentage of total haemoglobin
  Treatment period 1, N=11, 10 | 7.8 (1.3) | 7.4 (1.2)
  Treatment period 2, N=10, 12 | 7.6 (1.4) | 8.0 (1.0)

16. Secondary Outcome: Fasting Plasma Glucose
Description: Fasting plasma glucose (FPG) after each treatment period.
Time Frame: Week 16, week 32
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir First, Then Insulin NPH | Insulin NPH First, Then Insulin Detemir
Number analyzed (Participants) | 22 | 21
mmol/L
  Treatment period 1, N=12, 9 | 13.3 (5.8) | 10.5 (5.8)
  Treatment period 2, N=10, 12 | 9.1 (7.5) | 13.3 (5.2)

17. Secondary Outcome: Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes experienced in the study.
Time Frame: Weeks 0-32
Population: The safety analysis set included all randomised and exposed subjects.
Measure: Number; unit: episodes
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 23 | 23
episodes | 90 | 109

18. Secondary Outcome: Hypoglycaemic Episodes, Diurnal/Nocturnal
Description: Total number of hypoglycaemic episodes during the day (diurnal) and the night (nocturnal) experienced in the study.
Time Frame: Weeks 0-32
Population: The safety analysis set included all randomised and exposed subjects.
Measure: Number; unit: episodes
Arm/Group | Insulin Detemir | Insulin NPH
Number analyzed (Participants) | 23 | 23
episodes
  Diurnal | 62 | 60
  Nocturnal | 26 | 15
  Time of event not recorded | 2 | 34

ADVERSE EVENTS:
Time Frame: Adverse events were collected from July 2007 to July 2008.
Description: The safety analysis set included all randomised and exposed subjects.
Arm/Group | Insulin Detemir | Insulin NPH
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 7/23 | 4/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=23) | Insulin NPH (N=23)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Scratched eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Common cold (Infections and infestations) | 1 (1) | 1 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Viral gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Viral illness (Infections and infestations) | 0 (0) | 1 (1)
Slipped disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Panic attacks (Psychiatric disorders) | 1 (1) | 0 (0)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This open-label study was terminated prematurely due to 2 unplanned interim analyses having been performed. At this point, only 23 out of the planned 30 patients had been randomised into the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.